CLINICAL TRIAL: NCT05847218
Title: A Single-Dose Phase 1 Clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetics of RHN-001 in Healthy Adult Volunteers.
Brief Title: Phase 1 Clinical Trial of RHN-001 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RH Nanopharmaceuticals (Industry)
Collaborators: Center for Bioequivalence Studies and Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CB-046-RHN(S)-2021
Record Dates: First submitted 2023-03-22; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Safety; Tolerability; Pharmacokinetics
Keywords: Phase 1 study; Anti inflammatory; healthy volunteers

STUDY DESIGN:
Intervention Model Description: The study is planned to be conducted in Two Phases (Cohort A and Cohort B). The first phase will be carried out in two Cohorts i.e., single oral dose of investigational drug 750 mg or placebo under fasting (Cohort A1) and single oral dose of investigational drug 750 mg or placebo under fed conditions (Cohort A2). The second phase of the study will also be carried out in two cohorts i.e., single oral dose of 1500 mg or placebo under fasting (Cohort B1) and single oral dose of 1500 mg or placebo under fed conditions (Cohort B2). The second phase of the study will be carried out after the safety assessments of period one.
  Blood and urine samples will be collected from volunteers till 24 hours post dose in each Cohort for pharmacokinetic assessment of the drug and its active metabolites.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1 (750mg RHN-001 or Placebo) in fasting state (Experimental): Eligible 16 subjects will be randomized in Cohort A1 (n=16; 12 active: 4 Placebo) and fast for at least 10 hours on check-in day after dinner till 4 hours after they receive the investigational product (RHN-001 750mg caplet) or placebo at the study site on the morning of Day 2 of the study.
  Interventions: Drug: RHN-001 (one tablet 750mg)
- Cohort A2 (750mg RHN-001 or Placebo) in fed state (Experimental): Eligible 16 subjects will be randomized in Cohort A2 (n=16; 12 active: 4 Placebo) and will receive the investigational product (RHN-001) or placebo on Day 2 (dosing day) within 30 minutes after a standard breakfast. All subjects will undergo a 24-hour PK study during their stay at the clinical trial site.
  Interventions: Drug: RHN-001 (one tablet 750mg)
- Cohort B1 (1500mg RHN-001 or Placebo) in fasting state (Experimental): Eligible 16 subjects will be randomized in Cohort B1 (n=16; 12 active: 4 Placebo) and fast for at least 10 hours on check-in day after dinner till 4 hours after they receive the investigational product (RHN-001 1500mg caplet) or placebo at the study site on the morning of Day 2 of the study.
  Interventions: Drug: RHN-001 (750mg * 2 Tablets)
- Cohort B2 (1500mg RHN-001 or Placebo) in fed state (Experimental): Eligible 16 subjects will be randomized in Cohort B2 (n=16; 12 active: 4 Placebo) and will receive the investigational product (RHN-001) or placebo on Day 2 (dosing day) within 30 minutes after a standard breakfast. All subjects will undergo a 24-hour PK study during their stay at the clinical trial site.
  Interventions: Drug: RHN-001 (750mg * 2 Tablets)

INTERVENTIONS:
Drug: RHN-001 (one tablet 750mg) — Subjects in A1 and A2 will receive 750mg RHN-001 or matching placebo tablets in Fasted state and Fed states respectively with 240 mL ambient temperature water.
  Arms: Cohort A1 (750mg RHN-001 or Placebo) in fasting state; Cohort A2 (750mg RHN-001 or Placebo) in fed state
Drug: RHN-001 (750mg * 2 Tablets) — Subjects in B1 and B2 will receive 1500mg RHN-001 (750mg tablet) or matching placebo tablets in Fasted state and Fed states respectively with 240 mL ambient temperature water.
  Arms: Cohort B1 (1500mg RHN-001 or Placebo) in fasting state; Cohort B2 (1500mg RHN-001 or Placebo) in fed state

SUMMARY:
The goal of this clinical Trial is to assess the safety, tolerability and Pharmacokinetic profile of 750 mg single oral dose of RHN-001 and 1500 mg of RHN-001 administered orally in fasted and fed conditions in healthy adult volunteers.

DETAILED DESCRIPTION:
The study is planned to be conducted in Two Phases (Cohort A and Cohort B). The first phase will be carried out in two Cohorts i.e., a single oral dose of investigational drug 750 mg or placebo under fasting (Cohort A1) and a single oral dose of investigational drug 750 mg or placebo under fed conditions (Cohort A2).

The second phase of the study will also be carried out in two cohorts i.e., a single oral dose of 1500 mg or placebo under fasting (Cohort B1) and a single oral dose of 1500 mg or placebo under fed conditions (Cohort B2).

Blood samples will be obtained from the volunteers at different time-points i.e. 0.0 hour (before dosing), 15.0 minutes, 30.0 minutes, 1.0 hour, 2.0, 3.0, 4.0, 8.0, 12.0 and 24.0 hours post-dose in each cohort.

Urine samples (10 mL) for PK analysis will be collected after dosing for 24 hours whenever the subjects feel to urinate during their stay at the clinical trial site.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent obtained prior to any study-related procedures.
* Subject is a male/female with an age between 18 and 55 years of age, inclusive.
* Subject has a body mass index between 18 and 32 kg/m2, inclusive.
* Subject is judged to be in good health on the basis of medical history, complete physical examination, 12-lead electrocardiogram (ECG) and standard laboratory tests including complete hematology, blood chemistry, Lipid profile, Thyroid profile and urinalysis.
* Subject understands the procedures and agrees to participate in the study program.

Exclusion Criteria:

* Subject is under the age of legal consent, or is mentally or legally incapacitated.
* Subject has a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering RHN-001 to the subject.
* Subject has a recent history (10 years) of major cardiovascular, hepatic or renal disease.
* Subject has liver function tests abnormalities with elevated AST or ALT greater than or equal to 2 times upper limit of normal and/or elevated bilirubin greater than or equal to 2 times upper limit of normal.
* Subject has renal function tests abnormalities with serum creatinine greater than 1.8 g/dL.
* Subject has any clinically significant abnormal hematological values in the opinion of the principal investigator.
* Subject has abnormal serum concentrations of TSH, T3 or T4.
* Subject has clinically significant abnormalities at physical examination, ECG or laboratory tests carried out at screening.
* Subject has a history of psychiatric disorders, significant allergic conditions or known hypersensitivity to medications.
* Subject is positive on testing for hepatitis B surface antigen, hepatitis C antibody or HIV 1 or 2 antibodies or tested positive for COVID-19 on rapid antigen testing.
* Subject has donated blood within the 2 months before study drug administration.
* Subject has a history of alcohol or drug abuse within the past year.
* Subject used any over-the-counter drug during the 2 weeks prior to study drug administration (except occasional acetaminophen or vitamins).
* Subject is positive on urine drug screening for drugs of abuse (cannabinoids, cocaine, opiates, amphetamines, barbiturates, benzodiazepines).
* Subject tests positive for alcohol on Breath alcohol or urine screening.
* Subject smokes more than 5 cigarettes per day.
* Subject consumes caffeine more than 500 mg per day.
* Subjects unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study treatments.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability profile of SAD of RHN-001 | up to 24 hours post dose in each cohort
  Number of subjects with adverse events (AEs) (i.e., seriousness, severity, relationship to the study medication, outcome, duration, and management), vital signs, 12-lead electrocardiogram (ECGs), clinical laboratory parameters, weight, and physical examination.
Safety Endpoints of MAD of RHN-001 | up to 24 hours post dose in each cohort
  Number of subjects with adverse events (AEs) (i.e., seriousness, severity, relationship to the study medication, outcome, duration, and management), vital signs, 12-lead electrocardiogram (ECGs), clinical laboratory parameters, weight, and physical examination.

SECONDARY OUTCOMES:
maximum plasma concentration | up to 24 hours post dose
  maximum concentration of RHN-001 in plasma after dose in each cohort
Time to reach maximum plasma concentration | up to 24 hours post dose
  Time required for RHN-001 to reach maximum plasma concentration
AUC (Area under concentration vs time curve) | up to 24 hours post dose
  Area under the time versus plasma RHN-001 concentration curve

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Raza Shah, PhD, Principal Investigator — Center for bio-equivalence studies and clinical research, ICCBS, University of Karachi, Pakistan; Izhar Hasan, MD, PhD, Principal Investigator — RH Nanopharmaceuticals LLC, Princeton, NJ 088540
Locations (1):
- Center for Bioequivalence Studies and clinical research (CBSCR), ICCBS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
only de-identified individual participants data can be shared upon proper request to the sponsor.